CLINICAL TRIAL: NCT03721406
Title: The Pharmacokinetic of Ropivacaine in Patients Undergoing Ultrasound-guided Continuous Thoracic Paravertebral Block
Brief Title: Pharmacokinetic of Thoracic Paravertebral Ropivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Assoc Prof of Anaesthesiology, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROPICTPVB
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Open Thoracotomy
Keywords: ropivacaine; undergoing ultrasound guided thoracic paravertebral block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine (Other): * 25 ml single dose of 0.5% ropivacaine
  * continuous infusion of ropivacaine 0.2% with a constant infusion rate of 14 ml/h
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — ropivacaine administerd via thoracic paraveretebral catheter
  Other Names: thoracic paravertebral block

SUMMARY:
The study aims to investigate the pharmacokinetic of ropivacaine in patients undergoing ultrasound guided thoracic paravertebral block (TPVB) both after a single-bolus injection via the thoracic paravertebral catheter given before the start of surgery and after continuous thoracic paravertebral infusion that will start after the end of the procedure in order to achieve postoperative analgesia after open thoracotomy during the first 3 postoperative days

DETAILED DESCRIPTION:
Patients aged >18yrs, of ASA I-III undergoing open thoracotomy under combined ultrasound guided thoracic paravertebral block (TPVB) and general anesthesia will be enrolled in the study.

TPVB will be performed under ultrasound guidance on the side of the operation immediately after induction of anesthesia and patient intubation, with the patient in the lateral position at the T5 or T6 or T7 thoracic level using a Tuohy 17G needle and the catheter will be advanced 5 cm beyond the point of needle tip.

Dosage regimen Initially, after catheter placement and control, 0.5% ropivacaine is administered via the catheter in a 25 ml single dose, before the start of surgery.

After the end of surgery and patient awakening, the catheter will be connected with an electronic pump and the continuous infusion of ropivacaine 0.2% will start with a constant infusion rate of 14 ml/h for the first 3 postoperative days.

Postoperative pain will be assessed using the Visual Analogue Scale (VAS: 0-10). Postoperative analgesia will be managed with continuous PVB, and systemic administration of paracetamol (1 gr X 4 iv), tramadol (100 mg x 3 iv) and pregabalin (75 mg x 2 pos). Additionally, if VAS is ≥4-5 morphine (2.5 -5mg) will be administered subcutaneously as rescue analgesic drug (max 6 doses/day). In case of persistent pain (VAS > 4-5) despite the previously mentioned treatment measures, PCA morphine will be used.

Postoperative data include arterial blood pressure, heart rate, SpO2, VAS scores, clinical signs of local anesthetic toxicity during the first 3 postoperative days, specifically at 12, 24, 36, 48 and 72 postoperative hours.

Samples Serial blood samples from radial artery and central venous line will be collected at predefined time points, as following.

After the single-dose paravertebral injection Serial blood samples from radial artery will be collected at 5, 7.5, 10, 15, 20, end of surgery (min) Serial blood samples from central venous line will be collected at 1, 5, 7.5, 10, 15, 20, 40, 60, end of surgery (min)

After the initiation of continuous paravertebral infusion Serial blood samples from radial artery will be collected at 2.5, 7.5, 15, 30, 60 (min) and afterwards at 24, 48, 72 (hours) Serial blood samples from central venous line will be collected at 2.5, 10, 15, 30, 60 (min) and afterwards at 2, 6, 24, 48, 72 (hours)

Determination of ropivacaine plasma levels samples collected at regular intervals. All blood samples (2.5ml) will be placed into EDTA vacutainer tubes and immediately centrifuged (3,500rpm, 10min) after which the plasma will be Ropivacaine plasma levels will be measured in both arterial and venous blood removed. Plasma samples will be stored at -70 ° C until assayed. Bioassay of blood samples will be performed according to Good Laboratory Practice.

Measurement of ropivacaine plasma concentrations Quantification of total ropivacaine plasma levels in blood samples (sample volume 1mL) will be performed by high performance liquid chromatography (HPLC), using the method developed by Gaudreault F, Drolet P and Varin F (2009)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* ASA I-III
* Open thoracotomy

Exclusion Criteria:

* Patient refusal
* Age <18 years
* Morbid obesity
* Scoliosis
* Previous thoracotomy
* Empyema
* Drug allergy
* Severe systemic disease
* ASA > III
* Hypoalbuminemia
* Urgent surgery
* Reoperation during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
ropivacaine plasma levels | up to 72 postoperative hours after the initiation of continuous thoracic paravertebral infusion of ropivacaine
  Ropivacaine plasma levels in both arterial and venous blood samples collected at regular intervals

SECONDARY OUTCOMES:
Clinical signs of local anesthetic toxicity | Up to 72 hours after the initiation of continuous thoracic paravertebral infusion of ropivacaine
  Cardiac arrythmia on ECG

OTHER OUTCOMES:
VAS scores | up to 72 postoperative hours after the initiation of continuous thoracic paravertebral infusion of ropivacaine
  Postoperative pain will be assessed using the Visual Analogue Scale (0-10cm, 0=no pain, 10=the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi K Matsota, Prof, Principal Investigator — 2nd Department of Anaesthesiology, "Attikon" University Hospital, Athens
Locations (2):
- Greece (2):
  - 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica
  - Paraskevi K Matsota, Athens, Other

IPD SHARING:
Plan to Share IPD: No